CLINICAL TRIAL: NCT02743351
Title: A Phase 1, Non-Randomized, Open-Label/Phase 2, Randomized, Blinded Study of ProTmune™ (ex Vivo Programmed Mobilized Peripheral Blood Cells) Versus Non-Programmed Mobilized Peripheral Blood Cells for Allogeneic Hematopoietic Cell Transplantation in Adult Subjects With Hematologic Malignancies
Brief Title: Study of ProTmune for Allogeneic HCT in Adult Patients With Hematologic Malignancies
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Fate Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: PT-001
Record Dates: First submitted 2016-02-09; First posted 2016-04-19 (Estimated); Results first posted 2023-02-08 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2022-12

CONDITIONS: Hematologic Malignancies; Acute Myeloid Leukemia; Acute Lymphoblastic Leukemia; Myelodysplastic Syndromes; Chronic Myelogenous Leukemia; Acute Graft-versus-host Disease
Keywords: Cell Transplants; Hematopoietic Cell Transplant; HCT; Hematologic Malignancies; Hematologic Malignancy; Acute Myeloid Leukemia; Acute Lymphoblastic Leukemia; ALL; AML; Myelodysplastic Syndrome; MDS; Allogeneic; CML; Stem Cell Transplant; Transplant; aGvHD; Acute graft-versus-host Disease; cGvHD; Chronic graft-versus-host Disease
MeSH Terms: conditions — Hematologic Neoplasms; Leukemia, Myeloid, Acute; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Myelodysplastic Syndromes; Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Bronchiolitis Obliterans Syndrome

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ProTmune (Experimental): Conditioning regimen consisting of one of the following five preparative regimens: fludarabine and busulfan (FluBu4); busulfan (Bu) and cyclophosphamide (Cy); Cy and >or=12 Gy total body irradiation (TBI); TBI and etoposide; or fludarabine and melphalan (FluMel 140).
  Subjects will receive mPB cells from an available 8/8 HLA-A, -B, -C, and -DRB1-matched unrelated peripheral blood cell donor that were programmed ex vivo with ProTmune.
  Interventions: Biological: ProTmune
- Control Arm (Active Comparator): Conditioning regimen consisting of one of the following five preparative regimens: fludarabine and busulfan (FluBu4); busulfan (Bu) and cyclophosphamide (Cy); Cy and >or=12 Gy total body irradiation (TBI); TBI and etoposide; or fludarabine and melphalan (FluMel 140).
  Subjects will receive unmanipulated mPB cells from an available 8/8 HLA-A, -B, -C, and -DRB1-matched unrelated peripheral blood cell donor.
  Interventions: Biological: Control Arm

INTERVENTIONS:
Biological: ProTmune — Ex-vivo, programmed mobilized peripheral blood (mPB) cells
  Arms: ProTmune
Biological: Control Arm — Untreated mobilized peripheral blood (mPB) cells
  Arms: Control Arm

SUMMARY:
This study is a Phase 1, non-randomized, open-label/Phase 2 randomized, blinded study of ProTmune (ex vivo programmed mobilized peripheral blood cells) versus non-programmed mobilized peripheral blood cells for allogeneic hematopoietic cell transplantation (HCT) in adult subjects aged 18 years and older with hematologic malignancies. A total of 88 study subjects were treated in the trial at approximately 15 centers in the US.

ELIGIBILITY:
Key Inclusion Criteria:

1. Male and female patients aged 18 years and older, inclusive;
2. Patients must have a hematologic malignancy for which allogeneic hematopoietic peripheral blood cell transplantation is deemed clinically appropriate.

   Eligible diseases and stages include the following:
   1. Acute myeloid leukemia
   2. Acute lymphoblastic leukemia, including T lymphoblastic lymphoma with a history of marrow involvement
   3. Myelodysplastic Syndrome
   4. Chronic myelogenous leukemia
3. Availability of a suitable 8/8 HLA-A, -B, -C, and -DRB1-matched unrelated mPB donor;
4. mBP donor collection that meets protocol specifications;
5. Adequate performance status, defined as Karnofsky score greater than or equal to 70%;
6. For female patients of childbearing potential, all of the following criteria must be met:

   * They are not pregnant (i.e., female patients must have a negative serum pregnancy test at screening);
   * They are not breastfeeding;
   * They do not plan to become pregnant during the study; and
   * They are using an effective method of contraception from screening to the end of the study, unless their sexual partner is surgically sterile.
7. For male patients, agreement to use condoms with spermicide during sexual intercourse from screening to the end of study; and
8. Willingness and ability to sign an IRB/IEC-approved ICF before performance of any study-specific procedures or tests and to comply with protocol visits, and study procedures.

Key Exclusion Criteria:

1. Phase 1 only: Known bone marrow fibrosis; Phase 2 only: Bone marrow fibrosis grade 3 (severe) or greater;
2. Positive serology for human immunodeficiency virus (HIV) or human T-cell lymphotropic virus (HTLV) at any time prior to enrollment;
3. Currently uncontrolled bacterial, viral, or fungal infection (progression of clinical symptoms despite therapy);
4. Prior autologous or allogeneic HCT;
5. Active malignancy, other than the one for which the allogeneic mPB transplant is being performed, within 12 months of enrollment, excluding superficial basal cell and carcinoma in situ cervical cancer;
6. Pulmonary disease, renal dysfunction, hepatic disease, cardiac disease, neurologic disease;
7. Participation in another clinical trial involving an investigational product within 30 days prior to screening; or
8. Any condition or therapy, which, in the opinion of the Investigator, might pose a risk to the patient or make participation in the study not in the best interest of the patient.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2016-12-20 (Actual); Primary Completion 2020-12-04 (Actual); Study Completion 2021-11-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Cooley, MD, Study Director — Fate Therapeutics
Locations (15):
- United States (15):
  - University of Alabama, Birmingham, Alabama
  - City of Hope, Duarte, California
  - University of California, San Diego (UCSD) Moores Cancer Center, San Diego, California
  - University of Chicago, Chicago, Illinois
  - Indiana Blood and Marrow Transplant, Indianapolis, Indiana
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - Weill Cornell Medicine, New York, New York
  - Jewish Hospital, Cincinnati, Ohio
  - The Ohio State University, Columbus, Ohio
  - Oregon Health & Science University, Portland, Oregon
  - Sarah Cannon Research Institute, Nashville, Tennessee
  - Texas Transplant Institute, San Antonio, Texas
  - Huntsman Cancer Institute (University of Utah), Salt Lake City, Utah
  - Virginia Commonwealth University, Richmond, Virginia

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Phase I ProTmune; Phase 2 ProTmune: ProTmune: Ex-vivo, programmed mobilized peripheral blood (mPB) cells
- Phase 2 Control: Control Arm: Untreated mobilized peripheral blood (mPB) cells
Period: Overall Study
Arm/Group | Phase I ProTmune | Phase 2 ProTmune | Phase 2 Control
Started | 7 | 45 | 44
Completed (Patients who completed study through day +100) | 7 | 35 | 36
Not Completed | 0 | 10 | 8

BASELINE CHARACTERISTICS:
Population: Intent-to-Treat population
Groups:
- Total: Total of all reporting groups
Arm/Group | Phase I ProTmune | Phase 2 ProTmune | Phase 2 Control | Total
Number analyzed (Participants) | 7 | 45 | 44 | 96
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.4 (12.35) | 52.4 (13.07) | 50.7 (15.10) | 51.9 (13.94)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 13 | 23 | 41
  Male | 2 | 32 | 21 | 55
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 3 | 3
  Not Hispanic or Latino | 7 | 45 | 41 | 93
  Unknown or Not Reported | 0 | 0 | 0 | 0
Time from initial diagnosis of primary disease (months) [Mean (Standard Deviation); unit: months] — Population: For Phase 2, one participant in each group (ProTmune and Control) diagnosis date was not available.
  months
    number analyzed (Participants) | 7 | 44 | 43 | 94
    (all) | 5.4 (1.3) | 7.3 (7.12) | 8.4 (12.39) | 7.6 (9.67)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Cumulative Incidence of Grade II to IV aGvHD Through Day +100 Based on Investigator Assessment
Description: Acute GvHD (aGvHD) is assessed by assigning the clinical stage for the target organs (skin, liver, and gut) along with assigning an overall grade based on the minimum degree of organ involvement required to confer that grade. Grade II is defined as Stage 1 skin, Stage 1 liver, or Stage 1 GI; Grade III is defined as any Stage 1-3 skin, and Stage 2-3 liver, or Stage 2-4 GI; Grade IV is defined as Stage 4 skin, or Stage 4 liver and any Stage GI. A higher overall grade indicates a more severe outcome. The cumulative incidence of CIBMTR Grade II to IV aGVHD through approximately 100 days following HCT is measured by the percentage of participants who experienced grade II to IV aGVHD. The cumulative incidence and the associated 95% confidence interval are estimated using a competing risk analysis with death and relapse without grade II-IV aGvHD as a competing risk.
Time Frame: 100 days post-HCT
Population: Modified intent-to-treat (mITT) population
  * Phase 1: All subjects who received ProTmune
  * Phase 2: All randomized subjects who received Investigational Product (ProTmune or Control mPB units)
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Phase I ProTmune: Subjects with an available 8/8 human leukocyte antigen (HLA)-A, -B, -C, and -DRB1-matched unrelated peripheral blood cell donor who received 1 unit of ProTmune ex vivo programmed mPB cells.
- Phase 2 ProTmune: Subjects with an available 8/8 HLA-A, -B, -C, and -DRB1-matched unrelated peripheral blood cell donor who were randomized to received 1 unit of ProTmune ex vivo programmed mPB cells.
- Phase 2 Control: Subjects with an available 8/8 HLA-A, -B, -C, and -DRB1-matched unrelated peripheral blood cell donor who were randomized to received 1 unit of unmanipulated mPB cells.
Arm/Group | Phase I ProTmune | Phase 2 ProTmune | Phase 2 Control
Number analyzed (Participants) | 7 | 40 | 41
percentage of participants | 42.9 [7.6 to 75.7] | 44.4 [28.1 to 59.5] | 24.9 [12.7 to 39.1]

2. Secondary Outcome: 1-year GvHD-free, Relapse-free Survival (GRFS)
Description: 1-year GvHD-free, relapse-free survival (GRFS) is a composite endpoint in which events included Grade III to IV aGvHD, cGvHD requiring systemic immunosuppressive therapy, relapse, or death from any cause. GRFS is defined as the time from HCT to the earlier of the dates of the first documented CIBMTR Grade III-IV aGvHD, first use of systemic immunosuppressive therapy for cGvHD, first documented relapse of the underlying malignancy, or death from any cause. Subjects who are alive with no documented events for Grade III-IV aGvHD, use of systemic immunosuppressive therapy for cGvHD, relapse, or death at the data cutoff will be censored at their last visit date or follow-up on or prior to the date of one-year study completion/early discontinuation. The Kaplan-Meier estimate of the median GRFS and the 95% CI are presented
Time Frame: 365 days post-HCT
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: GRFS days
Groups:
- Phase 2 Control Arm: Control Arm: Untreated mobilized peripheral blood (mPB) cells
Arm/Group | Phase I ProTmune | Phase 2 ProTmune | Phase 2 Control Arm
Number analyzed (Participants) | 7 | 40 | 41
GRFS days | 218.0 [37.0 to NA] — The upper limit of the 95% confidence interval is not estimable. | 209.0 [140.0 to 351.0] | 296.0 [238.0 to NA] — The upper limit of the 95% confidence interval is not estimable.

3. Secondary Outcome: Percentage of Subjects Alive Without Relapse and Without Moderate or Severe cGvHD at Day +365 - mITT Population
Description: Percentage of subjects alive without relapse and without moderate or severe cGvHD per NIH Consensus Criteria at Day +365
Time Frame: 365 days post-HCT
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Phase I ProTmune | Phase 2 ProTmune | Control Arm
Number analyzed (Participants) | 7 | 40 | 41
percentage of participants | 42.9 [9.9 to 81.6] | 65.0 [48.3 to 79.4] | 53.7 [37.4 to 69.3]

ADVERSE EVENTS:
Time Frame: From first dose of investigational product up to 730 days post-HCT
Description: Non-serious AEs were reported by the investigator from Day -10 through Day +365 post-HCT. All SAEs were reported by the investigator from Day -10 through +365; only those SAEs considered by the investigator to be related to investigational product/study procedure were reported up to Day +730 post-HCT. All-cause mortality and AE reporting are based on the safety population, defined as all subjects who received investigational product.
Groups:
- Phase I ProTmune: Subjects with an available 8/8 human leukocyte antigen (HLA)-A, -B, -C, and -DRB1-matched unrelated peripheral blood cell donor who received 1 unit of ProTmune ex vivo programmed mPB cells.
  Safety population includes all subjects who received IP. Subjects in the treatment group represent the actual treatment received, regardless of the treatment the subject was allocated to receive at randomization.
  All-cause mortality includes measure of all deaths, due to any cause, that occurred during the study in the Intent-to-treat (ITT) population, defined as all Phase 1 subjects who received ProTmune ex vivo programmed mPB cells.
- Phase 2 ProTmune: Subjects with an available 8/8 HLA-A, -B, -C, and -DRB1-matched unrelated peripheral blood cell donor who were randomized to received 1 unit of ProTmune ex vivo programmed mPB cells.
  Safety population includes all subjects who received IP (ProTmune or Control). Subjects in the treatment group represent the actual treatment received, regardless of the treatment the subject was allocated to receive at randomization.
  All-cause mortality includes measure of all deaths, due to any cause, that occurred during the study in the Intent-to-treat (ITT) population, defined as all subjects in the randomized treatment group, regardless of actual treatment received.
- Control Arm: Subjects with an available 8/8 HLA-A, -B, -C, and -DRB1-matched unrelated peripheral blood cell donor who were randomized to received 1 unit of unmanipulated mPB cells.
  Safety population includes all subjects who received IP (ProTmune or Control). Subjects in the treatment group represent the actual treatment received, regardless of the treatment the subject was allocated to receive at randomization.
  All-cause mortality includes measure of all deaths, due to any cause, that occurred during the study in the Intent-to-treat (ITT) population, defined as all subjects in the randomized treatment group, regardless of actual treatment received.
Arm/Group | Phase I ProTmune | Phase 2 ProTmune | Control Arm
All-Cause Mortality (participants affected / at risk) | 2/7 | 12/40 | 6/41
Serious Adverse Events (participants affected / at risk) | 3/7 | 24/40 | 20/41
Other Adverse Events (participants affected / at risk) | 7/7 | 40/40 | 41/41
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase I ProTmune (N=7) | Phase 2 ProTmune (N=40) | Control Arm (N=41)
Acute GVHD in intestine (Immune system disorders) | 2 | 9 | 2
Acute GVHD in liver (Immune system disorders) | 0 | 2 | 0
Acute GVHD in skin (Immune system disorders) | 0 | 1 | 0
Chronic GVHD in intestine (Immune system disorders) | 1 | 0 | 2
Chronic GVHD in liver (Immune system disorders) | 0 | 1 | 0
Engraftment syndrome (Immune system disorders) | 0 | 1 | 0
Staphylococcal bacteraemia (Infections and infestations) | 1 | 1 | 0
Cellulitis (Infections and infestations) | 0 | 1 | 0
Clostridium difficile colitis (Infections and infestations) | 0 | 1 | 0
Cytomegalovirus colitis (Infections and infestations) | 1 | 0 | 1
Device related infection (Infections and infestations) | 0 | 1 | 0
Enterobacter sepsis (Infections and infestations) | 1 | 0 | 0
Enterococcal infection (Infections and infestations) | 1 | 0 | 0
Escherichia bacteraemia (Infections and infestations) | 0 | 1 | 0
Klebsiella bacteraemia (Infections and infestations) | 1 | 0 | 0
Klebsiella infection (Infections and infestations) | 0 | 1 | 0
Meningoencephalitis herpetic (Infections and infestations) | 0 | 1 | 0
Parotitis (Infections and infestations) | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 1 | 1
Pneumonia fungal (Infections and infestations) | 0 | 1 | 0
Sepsis (Infections and infestations) | 0 | 1 | 0
Sinusitis fungal (Infections and infestations) | 0 | 1 | 0
Bacterial sepsis (Infections and infestations) | 0 | 0 | 1
Corona virus infection (Infections and infestations) | 0 | 0 | 1
Enterocolitis infectious (Infections and infestations) | 0 | 0 | 1
Gastroenteritis viral (Infections and infestations) | 0 | 0 | 1
Respiratory syncytial virus bronchiolitis (Infections and infestations) | 0 | 0 | 1
Serratia bacteraemia (Infections and infestations) | 0 | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 1 | 3 | 2
Calculus ureteric (Renal and urinary disorders) | 0 | 1 | 0
Renal colic (Renal and urinary disorders) | 0 | 1 | 0
Renal failure (Renal and urinary disorders) | 0 | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
Organising pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pyrexia (General disorders) | 0 | 3 | 1
Asthenia (General disorders) | 0 | 1 | 1
Multi-organ failure (General disorders) | 0 | 1 | 0
Acute myocardial infarction (Cardiac disorders) | 0 | 1 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 0 | 0
Supraventricular extrasystoles (Cardiac disorders) | 1 | 0 | 0
Atrioventricular block (Cardiac disorders) | 0 | 0 | 1
Pericardial effusion (Cardiac disorders) | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 0
Gastritis (Gastrointestinal disorders) | 0 | 1 | 0
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 1
Veno-occlusive liver disease (Hepatobiliary disorders) | 0 | 2 | 1
Cholecystitis acute (Hepatobiliary disorders) | 1 | 0 | 0
Hepatic cirrhosis (Hepatobiliary disorders) | 0 | 0 | 1
Hepatic failure (Hepatobiliary disorders) | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 0 | 1 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 1 | 0
Ejection fraction decreased (Investigations) | 0 | 1 | 0
Platelet count decreased (Investigations) | 0 | 1 | 0
Neutrophil count decreased (Investigations) | 0 | 0 | 2
Autoimmune encephalopathy (Nervous system disorders) | 0 | 1 | 0
Posterior reversible encephalopathy syndrome (Nervous system disorders) | 1 | 0 | 0
Seizure (Nervous system disorders) | 1 | 0 | 0
Somnolence (Nervous system disorders) | 0 | 1 | 0
Autonomic nervous system imbalance (Nervous system disorders) | 0 | 0 | 1
Encephalopathy (Nervous system disorders) | 0 | 0 | 1
Haemorrhage intracranial (Nervous system disorders) | 0 | 0 | 1
Myopathy (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 2 | 0
Jugular vein thrombosis (Vascular disorders) | 0 | 1 | 0
Hypotension (Vascular disorders) | 0 | 0 | 2
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 0
Haemolytic uraemic syndrome (Blood and lymphatic system disorders) | 0 | 0 | 1
Optic nerve disorder (Eye disorders) | 0 | 1 | 0
Engraft failure (Injury, poisoning and procedural complications) | 0 | 1 | 1
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 1
Failure to thrive (Metabolism and nutrition disorders) | 0 | 0 | 1
Mental status changes (Psychiatric disorders) | 0 | 1 | 1
Chronic graft-versus-host disease (Immune system disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Phase I ProTmune (N=7) | Phase 2 ProTmune (N=40) | Control Arm (N=41)
Stomatitis (Gastrointestinal disorders) | 4 | 19 | 22
Nausea (Gastrointestinal disorders) | 3 | 13 | 20
Diarrhoea (Gastrointestinal disorders) | 2 | 12 | 12
Haemorrhoids (Gastrointestinal disorders) | 1 | 6 | 3
Vomiting (Gastrointestinal disorders) | 2 | 5 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 6 | 6
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 5 | 6
Abdominal distension (Gastrointestinal disorders) | 0 | 3 | 3
Dysphagia (Gastrointestinal disorders) | 1 | 2 | 3
Flatulence (Gastrointestinal disorders) | 0 | 2 | 1
Oesophagitis (Gastrointestinal disorders) | 0 | 2 | 10
Oral pain (Gastrointestinal disorders) | 0 | 2 | 1
Colitis (Gastrointestinal disorders) | 0 | 1 | 3
Constipation (Gastrointestinal disorders) | 0 | 1 | 3
Dry mouth (Gastrointestinal disorders) | 0 | 1 | 4
Gastritis (Gastrointestinal disorders) | 1 | 0 | 0
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 3
Acute graft versus host disease in skin (Immune system disorders) | 3 | 21 | 15
Chronic graft versus host disease (Immune system disorders) | 4 | 18 | 16
Chronic graft versus host disease in skin (Immune system disorders) | 2 | 14 | 9
Chronic graft versus host disease in liver (Immune system disorders) | 3 | 9 | 9
Acute graft versus host disease in intestine (Immune system disorders) | 1 | 10 | 11
Chronic graft versus host disease in intestine (Immune system disorders) | 3 | 3 | 5
Acute graft versus host disease in liver (Immune system disorders) | 1 | 2 | 0
Anaemia (Blood and lymphatic system disorders) | 4 | 20 | 8
Febrile neutropenia (Blood and lymphatic system disorders) | 2 | 17 | 17
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 7 | 1
Neutropenia (Blood and lymphatic system disorders) | 0 | 2 | 1
Anaemia macrocytic (Blood and lymphatic system disorders) | 1 | 0 | 0
Pancytopenia (Blood and lymphatic system disorders) | 1 | 0 | 0
Thrombotic microangiopathy (Blood and lymphatic system disorders) | 1 | 0 | 0
Cytomegalovirus infection (Infections and infestations) | 3 | 4 | 2
Cytomegalovirus viraemia (Infections and infestations) | 2 | 4 | 5
Viraemia (Infections and infestations) | 0 | 6 | 3
Clostridium difficile colitis (Infections and infestations) | 0 | 5 | 0
Clostridium difficile infection (Infections and infestations) | 1 | 3 | 2
Upper respiratory tract infection (Infections and infestations) | 0 | 4 | 3
Epstein-Barr viraemia (Infections and infestations) | 0 | 3 | 1
Human herpesvirus 6 infection (Infections and infestations) | 1 | 2 | 1
Klebsiella bacteraemia (Infections and infestations) | 1 | 2 | 0
Pneumonia (Infections and infestations) | 1 | 2 | 0
Urinary tract infection (Infections and infestations) | 1 | 2 | 4
Urinary tract infection bacterial (Infections and infestations) | 1 | 2 | 0
Bacteraemia (Infections and infestations) | 1 | 1 | 1
Candida infection (Infections and infestations) | 0 | 2 | 0
Cellulitis (Infections and infestations) | 0 | 2 | 1
Escherichia bacteraemia (Infections and infestations) | 0 | 2 | 0
Rhinovirus infection (Infections and infestations) | 1 | 1 | 0
Skin infection (Infections and infestations) | 0 | 2 | 0
Bacterial disease carrier (Infections and infestations) | 1 | 0 | 0
Bacteroides bacteraemia (Infections and infestations) | 1 | 0 | 0
Bronchitis (Infections and infestations) | 1 | 0 | 0
Catheter site infection (Infections and infestations) | 1 | 0 | 0
Cytomegalovirus colitis (Infections and infestations) | 1 | 0 | 0
Enterocolitis bacterial (Infections and infestations) | 1 | 0 | 0
Localised infection (Infections and infestations) | 1 | 0 | 0
Oral candidiasis (Infections and infestations) | 0 | 1 | 5
Parainfluenzae virus infection (Infections and infestations) | 1 | 0 | 0
Staphylococcal bacteraemia (Infections and infestations) | 1 | 0 | 2
Urinary tract infection viral (Infections and infestations) | 0 | 0 | 3
Fatigue (General disorders) | 3 | 13 | 18
Mucosal inflammation (General disorders) | 2 | 10 | 6
Oedema peripheral (General disorders) | 1 | 7 | 3
Pyrexia (General disorders) | 1 | 3 | 1
Generalised oedema (General disorders) | 1 | 1 | 0
Non-cardiac chest pain (General disorders) | 0 | 2 | 1
Decreased appetite (Metabolism and nutrition disorders) | 1 | 8 | 12
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 8 | 3
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 5 | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 4 | 2
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 4 | 6
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 4 | 9
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 2 | 2
Hypernatraemia (Metabolism and nutrition disorders) | 1 | 1 | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 2 | 3
Metabolic acidosis (Metabolism and nutrition disorders) | 1 | 1 | 0
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 | 1 | 4
Platelet count decreased (Investigations) | 4 | 16 | 13
Neutrophil count decreased (Investigations) | 4 | 13 | 9
White blood cell count decreased (Investigations) | 3 | 10 | 8
Alanine aminotransferase increased (Investigations) | 1 | 6 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 4 | 0
Blood bilirubin increased (Investigations) | 0 | 4 | 3
International normalised ratio increased (Investigations) | 0 | 4 | 0
Blood creatinine increased (Investigations) | 1 | 1 | 4
Weight decreased (Investigations) | 1 | 1 | 5
Electrocardiogram QT prolonged (Investigations) | 1 | 0 | 0
Hepatic enzyme increased (Investigations) | 1 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 | 4 | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 4
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 1
Laryngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 2
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Hypertension (Vascular disorders) | 4 | 9 | 14
Deep vein thrombosis (Vascular disorders) | 1 | 3 | 0
Embolism (Vascular disorders) | 0 | 4 | 0
Hypotension (Vascular disorders) | 0 | 3 | 1
Infusion related reaction (Injury, poisoning and procedural complications) | 2 | 11 | 8
Allergic transfusion reaction (Injury, poisoning and procedural complications) | 1 | 1 | 1
Procedural hypertension (Injury, poisoning and procedural complications) | 0 | 2 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 0
Laceration (Injury, poisoning and procedural complications) | 1 | 0 | 0
Dysgeusia (Nervous system disorders) | 4 | 5 | 6
Headache (Nervous system disorders) | 0 | 5 | 4
Encephalopathy (Nervous system disorders) | 1 | 2 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 1 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 5 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 5 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 3 | 4
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 2 | 2
Myopathy (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Tendonitis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 5
Acute kidney injury (Renal and urinary disorders) | 2 | 7 | 9
Azotaemia (Renal and urinary disorders) | 0 | 2 | 0
Urinary tract pain (Renal and urinary disorders) | 1 | 1 | 0
Bladder spasm (Renal and urinary disorders) | 1 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 5 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 2 | 1
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 2
Confusional state (Psychiatric disorders) | 1 | 4 | 1
Insomnia (Psychiatric disorders) | 0 | 4 | 5
Agitation (Psychiatric disorders) | 0 | 2 | 2
Anxiety (Psychiatric disorders) | 0 | 2 | 0
Delirium (Psychiatric disorders) | 1 | 0 | 2
Atrial fibrillation (Cardiac disorders) | 1 | 3 | 3
Sinus tachycardia (Cardiac disorders) | 0 | 2 | 1
Dry eye (Eye disorders) | 0 | 2 | 0
Vision blurred (Eye disorders) | 0 | 2 | 1
Cholecystitis (Hepatobiliary disorders) | 0 | 2 | 0
Cholecystitis acute (Hepatobiliary disorders) | 1 | 0 | 0
Hyperparathyroidism (Endocrine disorders) | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (3):
  • Study Protocol (2019-04-01): https://cdn.clinicaltrials.gov/large-docs/51/NCT02743351/Prot_000.pdf
  • Statistical Analysis Plan (2021-02-17): https://cdn.clinicaltrials.gov/large-docs/51/NCT02743351/SAP_001.pdf
  • Informed Consent Form (2019-03-29): https://cdn.clinicaltrials.gov/large-docs/51/NCT02743351/ICF_002.pdf